CLINICAL TRIAL: NCT00392340
Title: An Open-Label, Multicentre, Phase II Study of TVD as Treatment for Children With Stage 4 Neuroblastoma Failing to Respond to First-Line Treatment According to HR-NBL-01/ E-SIOP [Topotecan-Vincristine-Doxorubicin in Children With Stage 4 Neuroblastoma Failing to Respond to COJEC (TVD)]
Brief Title: Topotecan, Vincristine, and Doxorubicin in Treating Young Patients With Refractory Stage 4 Neuroblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000508641; CCLG-NB-2006-05; EUDRACT-2005-000915-80; EU-20641
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma; disseminated neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Doxorubicin; Topotecan; Vincristine

INTERVENTIONS:
Biological: filgrastim
Drug: doxorubicin hydrochloride
Drug: topotecan hydrochloride
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, vincristine, and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving topotecan together with vincristine and doxorubicin works in treating young patients with refractory stage 4 neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess whether treatment with topotecan hydrochloride, vincristine, and doxorubicin hydrochloride can achieve a satisfactory response rate in pediatric patients with stage 4 neuroblastoma that failed to respond to rapid first-line treatment.

Secondary

* Determine time to progression in these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter, open-label study.

Patients receive topotecan hydrochloride IV over 30 minutes on days 1-5 and vincristine IV continuously and doxorubicin hydrochloride IV continuously over 48 hours on days 5 and 6. Patients also receive filgrastim (G-CSF) subcutaneously beginning on day 9 and continuing until blood counts recover. Treatment repeats every 21-28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve partial response (PR) after two courses of treatment receive an additional two courses. Patients who achieve complete response or very good PR are treated according to the standard therapy in protocol SIOP-EUROPE- HR-NBL-1. Patients who fail to achieve PR after 2 courses receive further treatment at the physician's discretion.

Patients are followed periodically for at least 3 years.

PROJECTED ACCRUAL: A total of 63 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage 4 neuroblastoma
* Failed to achieve adequate metastatic partial response after first-line therapy while enrolled on protocol SIOP-EUROPE-HR-NBL-1

PATIENT CHARACTERISTICS:

* Neutrophil count > 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.36 mg/dL
* Bilirubin ≤ 2.92 mg/dL
* AST and ALT < 2.5 times upper limit of normal
* Glomerular filtration rate ≥ 60 mL/min
* Normal cardiac function on echocardiography
* No severe organ dysfunction
* No active hepatitis C or hepatitis B virus positivity
* No HIV infection

PRIOR CONCURRENT THERAPY:

* No anti-tumor chemotherapy within the past 10 days
* No radiotherapy within the past 30 days
* No other investigational drugs within the past 30 days
* No prior doxorubicin hydrochloride

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (complete or partial) > 50% after 2 courses of topotecan hydrochloride, vincristine, and doxorubicin hydrochloride

SECONDARY OUTCOMES:
Progression-free survival at the time of local progression or relapse, progression of pre-existing metastases, metastatic relapse, second primary malignancy, or death from any cause
Toxicity and incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Guy Makin, MD, PhD, Study Chair — Royal Manchester Children's Hospital
Locations (11):
- United Kingdom (11):
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland